CLINICAL TRIAL: NCT03728647
Title: Multimedia Education on Knowledge, Injection Skill, Insulin Injection Self-efficacy, Injection Performance Rate, Educational Satisfaction, Nursing Hours, and Biophysical Indicators
Brief Title: The Effectiveness of Multimedia Education for Patients With Type 2 Diabe Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KMUH-IRB-20130146
Record Dates: First submitted 2018-10-28; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus; Insulin; Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: This study used a randomized repeated-measures experimental design. The experimental group received a multimedia health education program and the control group received a regular health education program.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multimedia health education (Experimental): The program (flat touch computer) consisted of knowledge and technology levels. Knowledge: diabetic introduction, treatment, management of hyper- and hypoglycemia, complications, and experience sharing of insulin injection by a patient group. Technology: steps of insulin injection skills and complete technology demonstration . The program contents were organized using a unit-based piecemeal teaching approach. Participants could adjust their learning pace according to individual situations and could practice injection skills using an injection mold during hospitalization. A diabetes educator has assessed the learning outcome of each participant after intervention. At the day of discharge from hospital, each participant would acquire a copy of the multimedia health education compact disc.
  Interventions: Behavioral: multimedia health education
- regular health education (Active Comparator): The regular (traditional) education program (a diabetes educator) consisted of knowledge and technology levels. Knowledge: diabetic introduction, treatment, management of hyper- and hypoglycemia, and complications. Technology: steps of insulin injection skills and complete technology demonstration.
  Interventions: Behavioral: regular health education

INTERVENTIONS:
Behavioral: multimedia health education — The program (flat touch computer) consisted of knowledge and technology levels. Knowledge: diabetic introduction, treatment, management of hyper- and hypoglycemia, complications, and experience sharing of insulin injection by a patient group. Technology: steps of insulin injection skills and complete technology demonstration . The program contents were organized using a unit-based piecemeal teaching approach. Participants could adjust their learning pace according to individual situations and could practice injection skills using an injection mold during hospitalization. A diabetes educator has assessed the learning outcome of each participant after intervention. At the day of discharge from hospital, each participant would acquire a copy of the multimedia health education compact disc.
  Arms: multimedia health education
Behavioral: regular health education — The traditional education program (a diabetes educator) consisted of knowledge and technology levels. Knowledge: diabetic introduction, treatment, management of hyper- and hypoglycemia, and complications. Technology: steps of insulin injection skills and complete technology demonstration.
  Arms: regular health education

SUMMARY:
A total of 72 type 2 diabetes who began insulin therapy using a pen injector participated in this study. The experimental (n = 36) and control (n = 36) groups received multimedia and regular health education program. Four structured questionnaires were used, and videotapes were applied to demonstrate injection skills.

DETAILED DESCRIPTION:
To explore the effectiveness of two types health education on knowledge in diabetes and insulin injection, skills in insulin injection, self-efficacy in insulin injection, injection performance rate, satisfaction with health education,nursing hours, and biophysical indicators among the type 2 diabetes who began insulin therapy using a pen injector.With a repeated measures experimental study design, a total of 72 type 2 diabetes who began insulin therapy using a pen injector participated in this study. The experimental (n = 36) and control (n = 36) groups received multimedia and regular health education program. Four structured questionnaires were used, and videotapes were applied to demonstrate injection skills.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 2 diabetes.
2. First received insulin injection with Lantus, Levemir or Novomix.
3. Ability to communicate in Mandarin or Taiwanese.
4. Ability to self-inject insulin.

Exclusion Criteria:

1. Cognitive impairment or dementia, inability to manage self-care.
2. Severe or unstable medical conditions.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-08-16 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2014-08-31 (Actual)

PRIMARY OUTCOMES:
diabetes and insulin injection related knowledge scale | Change from Baseline diabetes and insulin injection related knowledge to the thirteenth week after discharge from hospital
  The 20-item diabetes and insulin injection related knowledge scale consists of 4 domains: brief introduction to diabetes, precautions for diabetes medications and insulin injection, management of hyper- and hypoglycemia, and complications of diabetes. Total scores ranged from 0 to 20. Higher scores represent a better outcome.
insulin injection skills scale | Change from Baseline insulin injection skills to the thirteenth week after discharge from hospital
  The insulin injection skills scale was rated by a certified diabetes educator according to each participant's performance on the 12 steps of operating a prefilled pen injector (12 items; scores ranged from 0 to 12) and the 10 steps of operating a disposable pen injector (10 items; scores ranged from 0 to 10 ). Participants scored 1 point for each correct operation and 0 points for each incorrect operation. Higher scores represent a better outcome.
self-efficacy in insulin injection scale | Change from Baseline self-efficacy in insulin injection to the thirteenth week after discharge from hospital
  The 10-item self-efficacy in insulin injection scale was modified based on the General Self-Efficacy Scale. Total scores ranged from 10 to 50. Higher scores represent a better outcome.
The health education satisfaction scale | Change from the day prior to discharge satisfaction with health education to the thirteenth week after discharge from hospital
  The 10 items health education satisfaction scale consisted of 10 items, with total scores ranging from 10 to 50. Higher scores represent a better outcome.
nursing hours | Through intervention to the day prior to discharge from hospital, an average of 1 week
  The nursing hours were calculated by adding up the total time spent by the diabetes educator instructing each participant to perform insulin injection.

SECONDARY OUTCOMES:
glycated hemoglobin(HbA1C) | Change from Baseline HbA1C to the thirteenth week after discharge from hospital
  Record the concentration of HbA1C (%) from the lab data in medical record
blood creatinine | Change from Baseline blood creatinine to the thirteenth week after discharge from hospital
  Record the concentration of blood creatinine (mg/dl) from the lab data in medical record
insulin performance rate | Change from the first week after discharge insulin performance rate from hospital to the thirteenth week after discharge
  The rate of insulin injection at home

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chuan Huang, PHD, Study Director — National Tainan Junior College of Nursing

IPD SHARING:
Plan to Share IPD: No